CLINICAL TRIAL: NCT01485419
Title: Characterization of the Early Sex Hormone Milieu Post Injury and Relationship With Resuscitation Requirements and Coagulopathy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jason Sperry, Assistant Professor of Surgery and Critical Care, University of Pittsburgh
Other Study IDs: NTI early sex hormone trial
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Traumatic Injury
Keywords: Sex hormones; Testosterone; Estradiol
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Traumatic injury is a major public health problem with an immense societal cost. Despite improvements in trauma management, patients continue to suffer significant morbidity and mortality. Evidence suggests that males and females tolerate severe injury differently with a greater protection afforded to females. Determining the mechanisms responsible for these sex-based outcome differences after injury, focusing specifically on the early sex-hormone environment post-injury, may allow those at highest risk for poor outcome to be predicted and promote interventions that can improve outcomes for all injured patients. The goal of this study is to determine if the early sex hormone environment soon after injury has effects on the intensity of the immune response, resuscitation and blood transfusion requirements, and important clinical outcomes including mortality, organ failure and infection, following significant injury.

ELIGIBILITY:
Inclusion Criteria:

Injury, ICU admission

Exclusion Criteria:

Isolated TBI, Admission beyond 6 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Injured patients requiring ICU admission who arrive within 6 hours of injury
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Multiple Organ Failure | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States